

| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| Туре | Version | | Document Identifier | Effective Date |
| eldo clinical doc | 1.0; CURRENT; Most-Recent | t; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | • |

#### **CONFIDENTIAL**

#### STATISTICAL ANALYSIS PLAN FOR PROTOCOL 207468

A Proof of Concept (POC) Clinical Study to Evaluate the appearance of fine lines and wrinkles on a Developmental Cosmetic Moisturising Cream in Healthy Subjects Presenting Visible Signs of Ageing.

#### **BIOSTATISTICS DEPARTMENT**

#### GLAXOSMITHKLINE CONSUMER HEALTHCARE

184 Liberty Corner

Warren, NJ





| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | • |

### **Table of Contents**

| Glossary4 | 4 |
|---------------------------------------------------|-----|
| 1 Introduction5 | 5 |
| 2 Objectives | 5 |
| 3 Study Design | 6 |
| 4 Sample Size Determination | 6 |
| 5 Data Considerations | 7 |
| 5.1 Analysis Populations | 7 |
| 5.2 Subgroups/Stratification | 3 |
| 5.3 Time Windows 8 | 3 |
| 5.4 Missing Data Handling | 3 |
| 6 Demographics and Baseline Characteristics | 3 |
| 6.1 Subject Disposition | 3 |
| 6.2 Demographics | 3 |
| 7 Treatment Compliance and Concomitant Medication | 18 |
| 9 | ) |
| 7.1 Treatment Compliance9 | ) |
| 7.2 Concomitant Medications9 | ) |
| 8 Analysis | 9 |
| 8.1 Primary Analysis9 | ) |
| 8.2 Secondary Analysis 1 | 10 |
| 9 Safety Analysis | 1 ( |
| 10 Interim Analysis | 1( |
| 11 Topline Summary 1 | 11 |
| 12 Changes to Planned Analysis 1 | |
| 13 References 1 | |
| Appendix 1 Study Schedule | |
| Appendix 2 List of Tables, Figures & Listings | |
| ADDUNA 4 LIST OF FADICS, FIGURES & LISTINGS | 4 ~ |



| Document Name | Statistical Analysis CCI | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

## Appendix 3 Templates for Tables, Figures & Listings ..... 17



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

## Glossary

| CI | Confidence Interval |
|--------|-------------------------------------------------|
| ITT | Intent-to-Treat |
| PP | Per Protocol |
| AE | Adverse Event |
| MedDRA | Medical Dictionary for Regulatory<br>Activities |
| TE | Treatment Emergent |
| TEWL | Transepidermal Water Loss |



| Document Name | Statistical Analysis CCI | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

#### 1 Introduction

This document describes the statistical methods and data presentations to be used in the summary and analysis of the final data from Protocol 207468.

## 2 Objectives

| Objectives | Endpoints |
|---|---|
| Primary | |
| Evaluation of wrinkle dimensions | DermaTOP parameter R <sub>a</sub> at 4 weeks. |
| (change from baseline) of test product | |
| compared to no treatment on the | |
| Periocular / Crow's Feet Area. | |
| Secondary | |
| Evaluation of wrinkle dimensions | DermaTOP parameter R <sub>a</sub> at 2 weeks and |
| (change from baseline) of test product | 4 weeks (positive control only) |
| and positive control compared to no | _ |
| treatment in the Periocular / Crow's Feet | DermaTOP parameters R <sub>z</sub> , S <sub>a</sub> and S <sub>tm</sub> at 2 |
| Area. | and 4 weeks |
| | Clinical Fitzpatrick Wrinkle Score at 2 |
| | and 4 weeks |
| Evaluation of skin moisturisation (change | Instrumental Corneometer values at 2 and |
| from baseline) of test product and | 4 weeks |
| positive control compared to no treatment | |
| on the Sub-ocular/ Cheek Area. | |
| Evaluation of texture (change from | Texture ranking at 4 weeks |
| baseline) of test product and positive | |
| control compared to no treatment on the | |
| full face. | |
| Evaluation of skin elasticity (change | Instrumental Cutometer parameters R5 |
| from baseline) of test product and | and R7 at 2 and 4 weeks |
| positive control compared to no treatment | |
| on the Sub-ocular/ Cheek Area. | 7 |
| Evaluation of skin barrier (change from | Instrumental Trans-Epidermal Water |
| baseline) of test product and positive | Loss (TEWL) values at 2 and 4 weeks |
| control compared to no treatment on the | |
| Sub-ocular/ Cheek Area. | |
| To evaluate the general safety of the | Assessment of frequency and severity of |
| study products | Adverse Events (AEs) |



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recen | t; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

#### 3 Study Design

- Evaluator-blind
- Single study centre
- Split-face design
- Healthy female subjects aged 30 to 65 with self-reported sensitive skin and visible signs of aging (visual wrinkles) on the face
- Study treatments: Positive- (Olay ProX Wrinkle Smoothing Cream) and Untreated-control
- Randomisation was to two of the 3 treatment arms (test product, positive control, no treatment) with treatment arm assignment further randomised to either the right side or left side of the face. Therefore, a subject was randomised to one of the 6 possible treatment groups:

| Right Side of Face | Left Side of Face |
|--------------------|-------------------|
| Test Product | Positive Control |
| Test Product | No Treatment |
| Positive Control | No Treatment |
| Positive Control | Test Product |
| No Treatment | Test Product |
| No Treatment | Positive Control |

#### 4 Sample Size Determination

Approximately 90 healthy subjects will be screened to randomise at least 72 subjects to ensure 66 subjects complete the entire study. This will ensure approximately 44 subjects per treatment arm (test product, positive control, no treatment) or 22 per treatment group (test product/no treatment, test product/positive control, positive control/no treatment).



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recer | nt; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | • |

The sample size is based on clinical considerations. With 40 subjects, a difference between test product and untreated in the change from baseline in R<sub>a</sub> of at least 46% of the magnitude of the within-subject standard deviation of the difference would be detectable at two-sided alpha=0.05 with approximately 80% power.

#### 5 Data Considerations

#### 5.1 Analysis Populations

- The 'Intent to treat' (ITT) population includes all subjects who are randomised into the study and have at least one post-baseline clinical assessment available. All efficacy analyses will be based on the ITT population.
- The Safety population will include all subjects with at least one product application to either side of the face. All safety analyses will be performed using the Safety population.
- The Per Protocol (PP) population will consist of the subset of ITT subjects which excludes those subjects with significant protocol deviations. Protocol deviations will be identified prior to database unblinding and will include, but not be limited to, non-compliance with the protocol or product application and use of prohibited concomitant medications. Confirmatory analyses of at least the primary efficacy endpoint of DermaTOP R<sub>a</sub> and key secondary objective relating to Fitzpatrick wrinkle score will be performed on the PP population.

Subjects with a protocol violation that is deemed to affect facial skin assessments after a specific timepoint will be part of the PP population, but will have their data excluded from the assessment at which the protocol violation occurred.

Violations that may lead to the exclusion of data for PP analysis include, but are not limited to, the following:

- Violation of inclusion or exclusion criteria at screening or baseline that may affect facial skin assessments.
- Non-compliance with assigned treatment regimen.
- Use of prohibited treatment or medication before or during the study,



| Document Name | Statistical Analysis CCI | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

which it is felt will affect facial skin assessments.

Violations will be documented in the Population Definitions document. The content of this document will be agreed upon between the Biostatistician and Clinical Development Director or designee prior to database lock and breaking of the study blind.

A PP analysis will be performed on the primary and key secondary objective if there is more than 10% difference in the number of subjects evaluable in any of the treatment groups for the ITT and PP populations.

#### 5.2 Subgroups/Stratification

There was no stratification in this study.

#### 5.3 Time Windows

All data will be accepted for analysis. Deviations from the scheduled nominal visit days are not expected. Any deviations will be noted in the deviation log and visits may be considered for exclusion from the Per Protocol population.

#### 5.4 Missing Data Handling

Missing data will not be imputed. Dropouts will be included in analyses up to the point of discontinuation.

#### **6** Demographics and Baseline Characteristics

#### 6.1 Subject Disposition

The number of subjects screened, enrolled, randomised and completing the study will be presented by treatment arm (i.e. test product, positive control, no treatment) and overall as well as in a separate summary, by treatment group (i.e. each right side of body/left side of body treatment combinations to which subjects were randomised) and overall using frequency counts and percentages.

#### 6.2 Demographics

Age will be summarized descriptively using means, medians and standard deviations. Race and Fitzpatrick skin type scores will be summarised using frequency counts and percentages.



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recei | nt; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

#### 7 Treatment Compliance and Concomitant Medications

#### 7.1 Treatment Compliance

All deviations associated with the application of either the test product or positive control or the preservation of the lack of treatment, if so assigned, to the relevant side of the face will be listed.

#### 7.2 Concomitant Medications

Any concomitant medication use will be listed.

#### 8 Analysis

The primary objective will be to evaluate the change from baseline in wrinkle dimensions in the crow's feet area for the test product compared to no treatment after 4 weeks of twice daily product application. Given that this is a POC study, the study will be considered a success if at least a trend in favour of the test product is observed. There will be no adjustment to the critical alpha level of 0.05 to account for inflation due to multiplicity. P-values resulting from inferential testing will be considered primarily as summary statistics.

#### 8.1 Primary Analysis

The primary endpoint of the study will be change from baseline in Derma TOP parameter  $R_a$  at 4 weeks.

Baseline and change from baseline in DermaTOP parameters R<sub>a</sub>, R<sub>z</sub>, S<sub>a</sub> and S<sub>tm</sub> will be summarised (N, mean, standard deviation, median, minimum and maximum) by treatment arm (test product, Olay ProX Wrinkle Smoothing Cream, no treatment) for each study visit (weeks 2 and 4). For each parameter, test product versus no treatment and positive control versus no treatment will be compared for the change from baseline at 2 weeks, and 4 weeks, using analysis of covariance (ANCOVA) with subject (random effect), treatment, and side of face as main effects and baseline value as covariate. This approach allows for the inclusion of data from all subjects treated with a given treatment arm (test product, positive control or no treatment) regardless of the treatment group (test product/no treatment, test product/positive control, positive control/no treatment) to which they were randomised to derive estimates of treatment effect.

If the assumption of normality is rejected, an appropriate transformation to the data



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recer | nt; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | • |

may be performed to facilitate the above method of analysis. Least square means from the ANCOVA model for the change from baseline will be presented for each treatment arm and pairwise treatment comparisons, together with the 95% confidence intervals. In the absence of an appropriate data transformation, non-parametric analyses may be performed. In the event of the use of non-parametric analysis, median differences will be presented, together with 95% confidence intervals based on the Hodges-Lehmann method.

#### 8.2 Secondary Analysis

The same presentation and analysis methods, as outlined above, will be performed using change from baseline for other parameters; DermaTOP parameters Rz,  $S_a$  and  $S_{tm}$ , clinical wrinkle assessment, TEWL values, Corneometer values and Cutometer parameters R5 and R7.

The texture assessment resulting from the ranking of photos will inherently be an assessment of change from baseline. As such, the data resulting from these rankings will be tabulated by treatment arm as proportions with baseline image better and Day 29 image better and analysed using a logistic regression with effects for treatment arm and side of face included in the model

#### 9 Safety Analysis

Treatment emergent AEs are defined as events that start on or after the first treatment date. Events occurring following the start of treatment which were also reported before treatment began with <u>no change in severity or causality</u> will however <u>not</u> be considered treatment emergent.

AEs will be tabulated according to the current version of the MedDRA. Frequencies and percentages will be presented by product group and overall, for each system organ class, and for each preferred term. Summaries of treatment-emergent AEs, treatment-related treatment-emergent AEs, AEs leading to discontinuation, and serious AEs will be completed.

#### 10 Interim Analysis

Not Applicable



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recei | nt; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

## 11 Topline Summary

The following tables will be produced for the topline summary:

| Table No. | Description |
|---|---|
| 9.1 | Subject Disposition by Treatment Group – All Screened Subjects |
| 9.3.1.1 | Summary of DermaTOP Parameter R <sub>a</sub> at 4 weeks – ITT Population |
| 9.3.1.2 | Analysis of DermaTOP Parameter R <sub>a</sub> – Change from baseline at 4 weeks – ITT Population |
| 9.4.1 | Treatment-Emergent Adverse Events – Safety Population |
| 9.4.2 | Treatment-Emergent Treatment-Related Adverse events – Safety Population |

## 12 Changes to Planned Analysis

There are no changes to the protocol-planned analyses.

#### 13 References

None



| Document Name | Statistical Analysis CC 207468.docx | | |
|---|---|---|---|
| eldo clinical doc | 1.0: CURRENT: Most-Recent: Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | 000002000020100 | 10 / Ipi 2017 10:01:20 |

## **Appendix 1 Study Schedule**



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-F | Recent; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

| | | | | - |
|---|---|---|---|---|
| Procedure/ Assessment | Visit 1<br>Day -3 | Visit 2 <sup>1</sup><br>Day 1 | Visit 3 <sup>1</sup> Day 15 (+/- 24 hrs) | Visit 4 <sup>1</sup> Day 29 (+/- 24 hrs) |
| | Screening / | Baseline | Week 2 | Week 4 |
| | Washout | Treatment | Treatment | Treatment |
| Informed consent | X | | | |
| Demographics | X | | | |
| Medical History | X | | | |
| Current / Concomitant medication | X | X | X | X |
| Adverse Events | | X | X | X |
| Fitzpatrick Skin Type Assessment (Appendix 2) | X | | | |
| Diary Review (Compliance) <sup>4</sup> | | X | X | X |
| Continued Eligibility | | X | X | X |
| Clinical Fitzpatrick Wrinkle Score in Periocular / | X | X | X | X |
| Crow's Feet Area (Appendix 3) <sup>3</sup> | Λ | Λ | Λ | Λ |
| Inclusion / Exclusion Criteria | X | X | | |
| Subject Eligibility <sup>6</sup> | X | X | | |
| Study Cleanser and Diary Dispensing | X | | | |
| Randomisation <sup>2</sup> | | X | | |
| USR- CliP High Resolution Images Left and Right Side of Face 3,5,7 | | X | | X |
| DermaTOP Measurement <sup>3</sup> Periocular / Crow's Feet Area | | X | X | X |
| TEWL Measurement <sup>3</sup> in Sub-ocular/ Cheek Area | | X | X | X |
| Corneometer Measurement <sup>3</sup> in Sub-ocular/ | | X | X | X |
| Cheek Area | | Λ | Λ | Λ |
| Cutometer Measurement <sup>3</sup> in Sub-ocular/ Cheek | | X | X | X |
| Area | | | Λ | Λ |
| Test Product(s) Dispensing | | X | | |
| Supervised Test Product Application | | X | X | |
| Test Product, Study Cleanser and Diary Return | | | | X |
| Subject Discharge from Study | | | | X |

- 1. On the day of site visit, subjects will be instructed to cleanse their face in the morning with tap water only and not to apply the test product or control. Measurements and assessments will be performed at least 12 hours after the last application of test products.
- 2. Subjects to be randomised to one of three treatment groups: test product/positive control, test product/no treatment or positive control/no treatment at the baseline visit.
- 3. Subjects will be acclimatized in a controlled environment (temperature 20-22°C, relative humidity between 40-60%) for a period of at least 30 minutes before the clinical and instrumental assessments are performed (EEMCO, 1997).
- 4. Diary to be reviewed by investigator or designee to confirm and encourage subject compliance.
- 5. At the end of the study, a blinded lay panel will assess all of the high resolution images for Texture by texture ranking (Appendix 4).
- 6. Inclusion criteria 7b to be reviewed at Screening and Baseline.
- 7. A 30 minute waiting time will occur in an acclimatized room after the USR-CliP High Resolution Images.



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recei | nt; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | |

## **Appendix 2 List of Tables, Figures & Listings**

In all outputs, the treatment labels and order for presentation in tables and listings is:

- 1) Moisturising Cream
- 2) Olay ProX Cream
- 3) No Treatment

| Table No. | Table Title (including population) | Standard | Template |
|---|---|---|---|
| 9.1.1 | Subject Disposition by Treatment Group – All Screened Subjects | X | |
| 9.1.2 | Subject Disposition by Treatment Arm – All Screened Subjects | X | |
| 9.2.1.1 | Demographics – ITT Population | X | |
| 9.2.1.2 | Demographics – Safety Population | X | |
| 9.2.1.3 | Demographics – PP Population (if needed) | X | |
| 9.3.1.1 | Summary of DermaTOP Parameter R <sub>a</sub> at 4 weeks – ITT Population | | Table 9.3.2.1 |
| 9.3.1.2 | Analysis of DermaTOP Parameter R <sub>a</sub> – Change from baseline at 4 weeks – ITT | | Table 9.3.2.2 |
| 9.3.1.3 | Summary of DermaTOP Parameters R <sub>a</sub> at 4 weeks – PP Population (if needed) | | Table 9.3.2.1 |
| 9.3.1.4 | Analysis of DermaTOP Parameter R <sub>a</sub> – Change from baseline at 4 weeks – PP Population (if needed) | | Table 9.3.2.2 |
| 9.3.1.3 | Summary of DermaTOP Parameters – ITT Population (except primary endpoint) | | Table 9.3.2.1 |
| 9.3.1.4 | Analysis of DermaTOP Parameters – Changes from baseline – ITT Population (except primary endpoint) | | Table 9.3.2.2 |
| 9.3.2.1 | Summary of TEWL – ITT Population | | Appendix 3 |



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Re | ecent; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | • |

| 9.3.2.2 | Analysis of TEWL – Changes from Baseline – ITT Population | | Appendix 3 |
|---|---|---|---|
| 9.3.3.1 | Summary of Corneometry – ITT Population | | Table 9.3.2.1 |
| 9.3.3.2 | Analysis of Corneometry – Changes from Baseline – ITT Population | | Table 9.3.2.2 |
| 9.3.4.1 | Summary of Cutometer Parameters – ITT Population | | Table 9.3.2.1 |
| 9.3.4.2 | Analysis of Cutometer Parameters – Changes from Baseline – ITT Population | | Table 9.3.2.2 |
| 9.3.5.1 | Summary of Fitzpatrick Wrinkle Assessment<br>Score – ITT Population | | Table 9.3.2.1 |
| 9.3.5.2 | Analysis of Fitzpatrick Wrinkle Assessment<br>Score – Changes from Baseline – ITT<br>Population | | Table 9.3.2.2 |
| 9.3.5.3 | Summary of Fitzpatrick Wrinkle Assessment<br>Score – PP Population | | Table 9.3.2.1 |
| 9.3.5.4 | Analysis of Fitzpatrick Wrinkle Assessment<br>Score – Changes from Baseline – PP<br>Population | | Table 9.3.2.2 |
| 9.3.6.1 | Summary of Texture Rankings Based on USR-CliP Images – ITT Population | | Appendix 3 |
| 9.3.6.2 | Analysis of Texture Rankings Based on USR-<br>CliP Images – Change from baseline – ITT<br>Population | | Appendix 3 |
| 9.4.1 | Treatment-Emergent Adverse Events – Safety<br>Population | X | |



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Re | cent; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | • |

| 9.4.2 | Treatment-Emergent Treatment-Related | X |
|---|---|---|
| | Adverse events – Safety Population | |
| 9.4.3 | Treatment-Emergent Adverse Events by<br>Severity – Safety Population | X |
| 9.4.4 | Treatment-Emergent Treatment-Related Adverse Events by Severity – Safety Population | X |

All listings to be generated are the standard set.



| Document Name | Statistical Analysis CC 207468.docx | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | 33332433420100 | |

## **Appendix 3 Templates for Tables, Figures & Listings**



| Document Name | Statistical Analysis CC 207468.docx | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | · |

Page x of y Program Run Date:xxxx

Table 9.3.2.1 Summary of TEWL ITT Population (N=xx)

| Timepoint | | Moisturising Cream | Olay ProX Cream | No Treatment |
|---|---|---|---|---|
| Baseline | N | XX | XX | XX |
| | Missing | XX | XX | XX |
| | Mean | X.XX | X.XX | X.XX |
| | SD | X.XXX | X.XXX | X.XXX |
| | 95%CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| Day 15 | N | XX | XX | XX |
| | Missing | XX | XX | XX |
| | Mean | X.XX | X.XX | X.XX |
| | SD | X.XXX | X.XXX | X.XXX |
| | 95%CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| Day 15 Change from Baseline | N | XX | XX | XX |
| | Missing | XX | XX | XX |
| | Mean | X.XX | X.XX | X.XX |
| | SD | X.XXX | X.XXX | X.XXX |
| | 95%CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| | LSMean (±SE) | X.XX (X.XXX) | X.XX (X.XXX) | X.XX (X.XXX) |
| Day 29 | N | XX | XX | XX |
| | Missing | XX | XX | XX |
| | Mean | X.XX | X.XX | X.XX |
| | SD | X.XXX | X.XXX | X.XXX |
| | 95%CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |



| Document Name | Statistical Analysis CC 207468.docx | | |
|---|---|---|---|
| eldo clinical doc | 1.0: CURRENT: Most-Recent: Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | 0000020000020100 | 107101 2017 10:01:20 |

| Day 29 Change from Baseline | N | XX | XX | XX |
|---|---|---|---|---|
| | Missing | XX | XX | XX |
| | Mean | X.XX | X.XX | X.XX |
| | SD | X.XXX | X.XXX | X.XXX |
| | 95%CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| | LSMean (±SE) | X.XX (X.XXX) | X.XX (X.XXX) | X.XX (X.XXX) |

An increase in TEWL shows damage to the skin barrier function.

Programmers Note: Same format for Tables 9.3.1.1, 9.3.1.3, 9.3.3.1, 9.3.4.1, 9.3.5.1 - Change the title, including adding the parameters as a BY group (Derma TOP has 4 parameters:  $R_a$ ,  $R_z$ ,  $S_a$  and  $S_{tm}$ , and Cutometer has 2 parameters: R5 and R7) to match protocol.

<sup>\*</sup> Baseline is measured prior to any test product application.

<sup>#</sup> LSMean and standard error (SE) derived from ANCOVA with subject as random effect, treatment arm and side of face as fixed effects, and baseline value as covariate.



| Document Name | Statistical Analysis CC 207468.docx | | |
|---|---|---|---|
| eldo clinical doc | 1.0: CURRENT: Most-Recent: Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | *************************************** | 10 / Ipi 2017 10.01.20 |

Page 1 of 2 Program Run Date:xxxx

## Table 9.3.2.2 Analysis of TEWL Change from Baseline ITT Population (N=xx)

| Timepoint | | Difference | 95% Confidence Interval for the | P-Value |
|---|---|---|---|---|
| | | | Difference | |
| Day 15 | Moisturising Cream vs. No Treatment | X.XX | X.XX, X.XX | X.XXX |
| | Olay ProX Cream vs No Treatment | X.XX | X.XX, X.XX | X.XXX |
| | Moisturising Cream vs Olay Prox Cream | X.XX | X.XX, X.XX | X.XXX |
| Day 29 | Moisturising Cream vs. No Treatment | X.XX | X.XX, X.XX | X.XXX |
| | Olay ProX Cream vs No Treatment | X.XX | X.XX, X.XX | X.XXX |
| | Moisturising Cream vs Olay Prox Cream | X.XX | X.XX, X.XX | X.XXX |

Difference is the first named treatment adjusted (LS) mean change from baseline minus the second named treatment adjusted mean change from baseline. Analysis model (ANCOVA) included subject as random effect, treatment arm and side of face as fixed effects, and baseline value as covariate.

PROGRAMMER'S NOTE: Same format for Tables 9.3.1.2, 9.3.1.4, 9.3.3.2, 9.3.4.2, 9.3.5.2 - Change the title, including adding the parameters as a BY group (DermaTOP has 4 parameters:  $R_a$ ,  $R_z$   $S_a$  and  $S_{tm}$  and Cutometer has 2 parameters: R5 and R7) to match protocol.



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-R | Recent; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | • |

Page x of y Program Run Date:xxxx

# Table 9.3.6.1 Summary of Texture Rankings Based on USR-CliP Images ITT Population (N=xx)

| Lay Reader ID | | Moisturising Cream | Olay ProX Cream | No Treatment |
|---|---|---|---|---|
| 1 | N | XX | XX | XX |
| | Missing | XX | XX | XX |
| | Proportion Day 29<br>better than Baseline | X.XX | X.XX | X.XX |
| 2 | N | XX | XX | XX |
| | Missing | XX | XX | XX |
| | Proportion Day 29<br>better than Baseline | X.XX | X.XX | X.XX |
| etc | | XX | XX | XX |
| 24 | N | XX | XX | XX |
| | Missing | XX | XX | XX |
| | Proportion Day 29<br>better than Baseline | X.XX | X.XX | X.XX |
| Total | N | XX | XX | XX |
| | Missing | XX | XX | XX |
| | Proportion Day 29 better than Baseline | X.XX | X.XX | X.XX |
| | 95%CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |



| Document Name | Statistical Analysis CC 207468.docx | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | 0000024000420100 | 10 7 pt 20 17 10.0 1.20 |

Page x of y Program Run Date:xxxx

# Table 9.3.6.2 Analysis of Texture Rankings Based on USR-CliP Images ITT Population (N=xx)

| Timepoint | Difference in Proportions of Day 29 | 95% Confidence Interval for the | P-Value |
|---|---|---|---|
| | Image Better than Baseline | Difference | |
| | X.XX | X.XX, X.XX | X.XXX |
| Moisturising Cream vs. No Treatment | | | |
| Olay ProX Cream vs No Treatment | X.XX | X.XX, X.XX | X.XXX |
| Moisturising Cream vs Olay ProX Cream | X.XX | X.XX, X.XX | X.XXX |

Difference is the first named treatment minus the second named treatment.

Analysis model (logistic regression) included treatment arm and side of face as fixed effects.



| Document Name | Statistical Analysis CC | 207468.docx | | |
|---|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Re | ecent; Effective | 090032d580d23463 | 10-Apr-2017 13:34:23 |
| Reason For Issue | Auto Issue | | | • |

## **SIGNATURE PAGE**

Statistical Analysis CCI 207468.docx

| Date | Signed By |
|---------------------------------------|------------------------|
| 10-Apr-2017 02:06:40 | PPD |
| Justification | Biostatistics Approval |
| Date | Signed By |
| 10-Apr-2017 13:34:16 | PPD |
| Justification | Approved |
| | <u> </u> |
| Date | Signed By |
| Y | |
| Justification | |
| Date | Signed By |
| Justification | |
| · | |
| Date | Signed By |
| Justification | |
| o accinemental | |
| Date | Signed By |
| Justification | |



| Document Name | SAP Amendment 207648.doc | | |
|---|---|---|---|
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580d54792 | 12-Jun-2017 07:04:24 |
| Reason For Issue | Auto Issue | | _ |

#### **CONFIDENTIAL**

## AMENDMENT TO STATISTICAL ANALYSIS PLAN FOR PROTOCOL 207468

A Proof of Concept (POC) Clinical Study to Evaluate the appearance of fine lines and wrinkles on a Developmental Cosmetic Moisturising Cream in Healthy Subjects

Presenting Visible Signs of Ageing.

Biostatistics Department GlaxoSmithKline Consumer Health

PPD (Statistician)



| Document Name | SAP Amendment 207648.doc | | |
|---|---|---|---|
| Туре | Version Document Identifier Effective Date | | Effective Date |
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580d54792 | 12-Jun-2017 07:04:24 |
| Reason For Issue | Auto Issue | | |

**Timing of Amendment:** ⊠ Before unblinding ☐ After unblinding

**Section: 6.1 Subject Disposition** 

Reason for amendment: Clarification of the extent of reporting.

**Original text:** The number of subjects screened, enrolled, randomized and completing the study will be presented by treatment arm (i.e. test product, positive control, no treatment) and overall as well as in a separate summary, by treatment group (i.e. each right side of body/left side of body treatment combinations to which subjects were randomized) and overall using frequency counts and percentages.

Amendment: The number of subjects screened, enrolled, randomized and completing the study will be presented by treatment combination arm (i.e the pair of treatments received. test product, positive control, no treatment) with no account being made for side specific combinations – hence 3 columns. and overall as well as in a separate summary, by treatment group (i.e. each right side of body/left side of body treatment combinations to which subjects were randomized) and overall using frequency counts and percentages.

**Section: 9 Safety Analysis** 

Reason for amendment: Reference to additional pre-unblind step of assigning application site(s) AE's to treatment at that site(s).

**Original text:** Treatment emergent AEs are defined as events that start on or after the first treatment date. Events occurring following the start of treatment which were also reported before treatment began with <u>no change in severity or causality</u> will however not be considered treatment emergent.

AEs will be tabulated according to the current version of the MedDRA. Frequencies and percentages will be presented by product group and overall, for each system organ class, and for each preferred term. Summaries of treatment-emergent AEs, treatment-related treatment-emergent AEs, AEs leading to discontinuation, and serious AEs will be completed.

**Amendment:** Treatment emergent AEs are defined as events that start on or after the first treatment date. Events occurring following the start of treatment which were also



| Document Name | SAP Amendment 207648.doc | | |
|---|---|---|---|
| eldo_clinical_doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580d54792 | 12-Jun-2017 07:04:24 |
| Reason For Issue | Auto Issue | | |

reported before treatment began with <u>no change in severity or causality</u> will however <u>not</u> be considered treatment emergent.

AEs will be tabulated according to the current version of the MedDRA. Frequencies and percentages will be presented by product group and overall, for each system organ class, and for each preferred term. Summaries of treatment-emergent AEs, treatment-related treatment-emergent AEs, AEs leading to discontinuation, and serious AEs will be completed.

A further step will take place pre-unblind to flag the AEs by application site if appropriate so that attribution to applied treatment is preserved. This will involve review of all application site AEs and addition of a flag to indicate which site(s) it is applicable to.



| Document Name | SAP Amendment 207648.doc | | |
|---|---|---|---|
| Туре | Version Document Identifier Effective Date | | Effective Date |
| eldo clinical doc | 1.0; CURRENT; Most-Recent; Effective | 090032d580d54792 | 12-Jun-2017 07:04:24 |
| Reason For Issue | Auto Issue | | · |

## **SIGNATURE PAGE**

## SAP Amendment 207648.doc

| 12-Jun-2017 06:39:36 | Signed By Approved Signed By PPD |
|------------------------|----------------------------------|
| Justification A | Approved Signed By |
| Date S | Signed By |
| Date S | |
| Date S | |
| | PPD |
| 12-Jun-2017 07:04:18 | |
| <b>Justification</b> E | Biostatistics Approval |
| Date S | Signed By |
| Justification | |
| Date S | Signed By |
| Justification | |
| Date S | Signed By |
| Justification | |
| Date S | Signed By |
| Justification | |